CLINICAL TRIAL: NCT03530969
Title: Geriatric Communication Skills Training Program for Oncology Clinicians to Improve Management of Care for Geriatrics Cancer Patients
Brief Title: Geriatric Communication Skills Training Program for Oncology Clinicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-183
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: GI Cancer; Lymphoma; GU Cancer; Bone Marrow Transplant
MeSH Terms: conditions — Gastrointestinal Neoplasms; Lymphoma | interventions — Surveys and Questionnaires; Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GI/GU/Lymphoma Oncologists (Experimental): Doctors specializing in treating gastrointestinal cancer (cancer of the stomach, pancreas, colon, etc.), genitourinary cancer (cancer of the genitals and urinary tract), and lymphoma (cancer affecting the blood and lymph nodes)
  Interventions: Behavioral: Self-Efficacy Assessment; Behavioral: UCLA Geriatrics Attitudes Scale; Behavioral: Course Evaluations
- Participants with GI/GU/Lymphoma Cancer (Active Comparator): Patients of the physicians in group 1
  Interventions: Behavioral: The Consultation and Relational Empathy (CARE) questionnaire; Behavioral: Consumer Assessment of Health Care Providers and Systems Program (CAHPS); Behavioral: Patient activation measure (PAM) scale
- Caregivers of Participants with GI/GU/Lymphoma Cancer (Active Comparator): Family members or caregivers of the patients in group 2
  Interventions: Behavioral: The Consultation and Relational Empathy (CARE) questionnaire; Behavioral: Consumer Assessment of Health Care Providers and Systems Program (CAHPS)

INTERVENTIONS:
Behavioral: Self-Efficacy Assessment — Health Care Professional's self-efficacy will be assessed by 12 ratings of self-reported confidence from (1) "strongly disagree" to (5) "strongly agree" in module-specific topics both before and after the training.
  Arms: GI/GU/Lymphoma Oncologists
Behavioral: UCLA Geriatrics Attitudes Scale — The UCLA Geriatrics Attitudes Scale is a 14-item scale developed to assess health care providers' attitudes toward older persons and caring for older patients.
  Other Names: Perceived Ageism
  Arms: GI/GU/Lymphoma Oncologists
Behavioral: Course Evaluations — The evaluation surveys for each of the three modules will contain fifteen statements assessing post-training attitudes regarding the skills learned and application of skills in oncology clinical practice, measured on a 5-point Likert scale.
  Arms: GI/GU/Lymphoma Oncologists
Behavioral: The Consultation and Relational Empathy (CARE) questionnaire — The Consultation and Relational Empathy (CARE) questionnaire is a 10-item self-report scale that measures a patient's satisfaction with how empathic their health care providers (HCP) was within a specific consultation.
  Other Names: Perceived Empathy
  Arms: Caregivers of Participants with GI/GU/Lymphoma Cancer; Participants with GI/GU/Lymphoma Cancer
Behavioral: Consumer Assessment of Health Care Providers and Systems Program (CAHPS) — Patients" perceptions of the quality of their interactions with their clinicians will be rated with 6 items from the Consumer Assessment of Health Care Providers and Systems Program (CAHPS)
  Other Names: Satisfaction with communication
  Arms: Caregivers of Participants with GI/GU/Lymphoma Cancer; Participants with GI/GU/Lymphoma Cancer
Behavioral: Patient activation measure (PAM) scale — The PAM scale contains 22 items that assess patient engagement in their care process.
  Other Names: Patient Activation.
  Arms: Participants with GI/GU/Lymphoma Cancer

SUMMARY:
The purpose of this study is to learn more about the effects of a training program designed to help doctors communicate better with older patients and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

Clinician Eligibility

* MSK medical oncology Health Care Professionals (HCP) - specifically identified as Attendings, fellows, or Advance Practice Professional (APP) - either a Nurse Practitioner (NP) or Physician Assistant (PA) from GI, GU Oncology, Lymphoma, Bone Marrow Transplant or Geriatrics Service (five services with a large number of geriatric patients)
* Willingness to be audio-recorded as per self-report
* Clinician has individual clinic consultations with patients in the target population: 65 years of age and over, English speaking, and patients who have had a new visit within the last 6 months.

Patient Eligibility

* MSK patients 65 years of age and over as per EMR
* English speaking as per EMR
* Being seen by one of the consented HCPs as per the HCP and/or electronic medical record (EMR)
* Willingness to be audio-recorded as per self-report
* Patient had their first visit with the clinician within the last 6 months

Caregiver Eligibility

* English speaking as per EMR
* Accompanying an MSK patient being seen by one of the consented HCPs as per the HCP and/or EMR

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of Health Care Provider (HCP) training | 8 weeks
  Measured by number of HCP successfully recruited for the training
Participants satisfaction with Health Care Provider (HCP) training | 1 week
  Self-reported measure of satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Smita Banerjee, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org